CLINICAL TRIAL: NCT04580433
Title: Effects of 16:8 Time-restricted Feeding on the Endocrine and Metabolic Profile in Overweight Women With Polycystic Ovary Syndrome
Brief Title: Time-restricted Feeding for Treating Polycystic Ovary Syndrome (PCOS)
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chunzhu Li (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Chunzhu Li, Clinical Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020161820
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Polycystic Ovary Syndrome; Overweight; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-Restricted Feeding (Experimental): Participants will receive 16:8 TRF.
  Interventions: Behavioral: Time-Restricted Feeding

INTERVENTIONS:
Behavioral: Time-Restricted Feeding — The trial consists of a 1-week baseline weight stabilization period followed by a 5-week TRF intervention period.
  Participants will be instructed to eat freely from 8 a.m. to 4 p.m. daily and fast from 4 p.m. to 8 a.m. the next day.

SUMMARY:
Intermittent fasting is an increasingly popular diet pattern of alternating eating and dieting.One particular form of intermittent fasting is the so-called time-restricted feeding (TRF). TRF allows for ad libitum feeding within a large window of time each day, and does not require any calorie counting. There is growing evidence that it can lose weight, reduce insulin resistance and improve cardiometabolic health. Polycystic ovary syndrome (PCOS) is the most common reproductive endocrine and metabolic disease affecting women of childbearing age. PCOS shows anovulation or oligoovulation, hyperandrogenemia and ovarian polycystic changes. Insulin resistance and obesity are common features of PCOS. Whether the TRF impacts women with PCOS is still unknown due to the paucity of data in this area. To explore the effects of TRF on the endocrine and metabolic profile in overweight women with PCOS, a 6-week single-arm trial, divided into 2 consecutive periods: (1) 1-week baseline period; and (2) 5-week TRF period, will be implemented.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years; BMI≥24kg/m2; Anovulation; Rott-PCOS.

Exclusion Criteria:

Taking weight loss or regulate hormone secretion medications in recent 6 months; The body weight fluctuated more than 5% in the past 3 months; Preparation for pregnancy, having been in pregnancy or lactation; Perimenopausal; Night-shift workers; Fasting more than 16 hours a day; Hypotension; Patients with other diseases (such as congenital adrenal hyperplasia, Cushing syndrome, androgen-secreting tumors, hyperprolactinemia, diabetes, thyroid diseases, severe serious cardiovascular, gastrointestinal, kidney or liver diseases); Alcohol intake more than 100g per week; Smoking within 3 months; Engaging in high-intensity exercise.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with PCOS.
Enrollment: 18 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 5-week intervention period
  Will be assessed by homeostasis model assessment-insulin resistance (HOMA-IR)
Sex hormone-binding globulin (nmol/L) | 5-week intervention period
Body Mass Index (BMI) (kg/m^2) | 5-week intervention period
  Weight (kg) and height (m) will be combined to report BMI
Waist-to-Hip Ratio (WHR) | 5-week intervention period
  Waist and hip will be combined to report WHR
Free androgen index (FAI) (%) | 5-week intervention period
Total testosterone (TT) (ng/mL) | 5-week intervention period
Area under the curve (AUC) for insulin | 5-week intervention period
  Insulin release test will be conducted
Area under the curve (AUC) for glucose | 5-week intervention period
  Glucose tolerance test will be conducted
Area under the curve (AUC) for insulin/Area under the curve (AUC) for glucose | 5-week intervention period
  Glucose tolerance test will be conducted
Fasting insulin (FINS) (mU/L) | 5-week intervention period
Fasting blood glucose (FBG) (mmol/L) | 5-week intervention period

SECONDARY OUTCOMES:
Dietary behavior | 5-week intervention period
  Measured by the Three Factor Eating Questionnaire Revised 21 Item (TFEQ-R21) questionnaire
Time to return to normal menstrual cycle | 5-week intervention period
Insulin-like growth factor 1 (IGF-1) (ng/mL) | 5-week intervention period
Body fat (kg) | 5-week intervention period
  Measured by InBody, a body composition analyzer
Body fat percentage (%) | 5-week intervention period
  Measured by InBody, a body composition analyzer
Visceral fat area (cm^2) | 5-week intervention period
  Measured by InBody, a body composition analyzer
Skeletal muscle content (kg) | 5-week intervention period
  Measured by InBody, a body composition analyzer
High-sensitivity C-reactive protein (hs-CRP) (mg/L) | 5-week intervention period
  A kind of inflammatory biomarker

OTHER OUTCOMES:
Luteinizing hormone (LH) (mIU/mL) | 5-week intervention period
Follicle-stimulating hormone (FSH) (mIU/mL) | 5-week intervention period
LH/FSH | 5-week intervention period
Uric acid (UA) (umol/L) | 5-week intervention period
Alanine aminotransferase (ALT) (U/L) | 5-week intervention period
Aspartate aminotransferase (AST) (U/L) | 5-week intervention period
Total cholesterol (TC) (mmol/L) | 5-week intervention period
Triglycerides (TG) (mmol/L) | 5-week intervention period
Low density lipoprotein-cholesterol (LDL-C) (mmol/L) | 5-week intervention period
Body weight (kg) | 5-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Bing He, phD, Principal Investigator — Shengjing Hospital; Chunzhu Li, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li C, Xing C, Zhang J, Zhao H, Shi W, He B. Eight-hour time-restricted feeding improves endocrine and metabolic profiles in women with anovulatory polycystic ovary syndrome. J Transl Med. 2021 Apr 13;19(1):148. doi: 10.1186/s12967-021-02817-2. PMID 33849562